CLINICAL TRIAL: NCT02297841
Title: Repeated Insult Patch Test of Personal Lubricants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ST-7554
Record Dates: First submitted 2014-11-17; First posted 2014-11-21 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-09

CONDITIONS: Erythema; Edema
MeSH Terms: conditions — Erythema; Edema

ARMS (1):
- Human Repeat Insult Patch Test (Experimental): Approximately 0.2ml of each intervention (Experimental: Novel lubricant Miami Fragrance, Experimental: Novel lubricant Miami no Fragrance, KY Liquid lubricant, Astroglide Gel lubricant) was applied to an occlusive patch and applied to participant's back.
  Interventions: Device: Experimental: Novel lubricant Miami Fragrance; Device: Experimental: Novel lubricant Miami no Fragrance; Device: KY Liquid lubricant; Device: Astroglide Gel lubricant

INTERVENTIONS:
Device: Experimental: Novel lubricant Miami Fragrance
Device: Experimental: Novel lubricant Miami no Fragrance
Device: KY Liquid lubricant
Device: Astroglide Gel lubricant

SUMMARY:
Determine the ability of the study material (personal lubricant) to cause sensitization by repeated topical application to the skin of humans under controlled patch test conditions.

ELIGIBILITY:
Inclusion Criteria:

* In general good health
* Free of any systemic or dermatologic disorder which, in the opinion of the investigative personnel, will interfere with the study results or increase the risk of adverse events
* Are of any skin type or race, providing the skin pigmentation will allow discernment of erythema
* Complete a medical screening procedure
* Read, understand, and sign an informed consent agreement

Exclusion Criteria:

* Have any visible skin disease at the study site which, in the opinion of the investigative personnel, will interfere with the evaluation
* Are receiving systemic or topical drugs or medication which, in the opinion of the investigative personnel, will interfere with the study results
* Have psoriasis and/or active atopic dermatitis/eczema.
* Are females who are pregnant, planning on getting pregnant during the study, or breast-feeding
* Have a known sensitivity for cosmetics, skin care products, topical drugs, or any other type of the products, as related to the material being evaluated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Human Repeat Insult Patch Test: Experimental: Human Repeat Insult Patch Test
  Approximately 0.2ml of each intervention (Experimental: Novel lubricant Miami Fragrance, Experimental: Novel lubricant Miami no Fragrance, KY Liquid lubricant, Astroglide Gel lubricant) was applied to an occlusive patch and applied to participant's back.
Period: Overall Study
Arm/Group | Human Repeat Insult Patch Test
Started | 209
Induction Phase | 209
Challenge Phase | 201
Completed | 201
Not Completed | 8
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 7

BASELINE CHARACTERISTICS:
Groups:
- HRIPT: Novel lubricant Miami w/ fragrance Novel lubricant Miami w/o fragrance 510(k) cleared and currently marketed personal lubricant 510(k) cleared and currently marketed personal lubricant
Arm/Group | HRIPT
Number analyzed (Participants) | 201
Age, Customized [Number; unit: participants]
  18-70 | 201
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Time Frame: 24, 48, and 72 hours after patch application
Measure: Number; unit: participants
Arm/Group | Human Repeat Insult Patch Test
Number analyzed (Participants) | 201
participants | 0

ADVERSE EVENTS:
Groups:
- HRIPT: Experimental: Novel lubricant Miami w/ frag Experimental: Novel Miami w/o frag KY Liquid lubricant Astroglide Gel lubricant
Arm/Group | HRIPT
Serious Adverse Events (participants affected / at risk) | 0/209
Other Adverse Events (participants affected / at risk) | 0/209

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Master service agreement and confidentiality agreement in place